CLINICAL TRIAL: NCT02650856
Title: Blood Loss Reduction After Total Knee Arthroplasty. A Comparison Between Topical Tranexamic Acid and Platelet Rich Plasma: Controlled Clinical Trial
Brief Title: Blood Loss Reduction After Total Knee Arthroplasty. Comparison Topical Tranexamic Acid vs Platelet Rich Plasma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, FELIX VILCHEZ CAVAZOS, Dr. med. José Félix Vilchez Cavazos, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OR15-007
Record Dates: First submitted 2015-12-29; First posted 2016-01-08 (Estimated); Results first posted 2020-02-27 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Osteoarthritis
Keywords: Blood loss; Tranexamic acid; Platelet rich plasma; Total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 Tranexamic acid (Experimental): A dosis of 2 gr of tranexamic acid (1000mg/10ml X-GEN pharmaceuticals inc.) diluted in 80ml of physiologic solution and will be divided in two applications.
  First application: 40ml of the solution previously prepared is applied over the surgical site and it will be left for five minutes then drained out completely by suction.
  Second application: The rest of 40ml of solution previously prepared is applied after placing the final TKR components (femoral, tibial and patellar), over the surgical site and leaving it without draining it by suction.
  Interventions: Drug: Group 1 Tranexamic Acid
- Group 2 Platelet rich plasma (Active Comparator): A final volumen of 16 ml of platelet rich plasma is obtained from the forearm vein of the patient and will be divided in two applications.
  First application: 8 ml of PRP are applied over the surgical site and are left for five minutes then drained out completely by suction.
  Second application: The rest of the 8 ml are applied after placing the final TKR cemented components (femoral, tibial and patellar), over the surgical site and leaving it without draining.
  Interventions: Biological: Group 2 Platelet rich plasma

INTERVENTIONS:
Drug: Group 1 Tranexamic Acid — 2 gr of tranexamic acid will be applied on the surgical site.
  Other Names: Topic Tranexamic Acid
  Arms: Group 1 Tranexamic acid
Biological: Group 2 Platelet rich plasma — 16ml of platelet rich plasma will be applied of the surgical site
  Other Names: PRP
  Arms: Group 2 Platelet rich plasma

SUMMARY:
The investigators will include patients who will be schedule for total knee arthroplasty with a diagnosis of osteoarthritis. The patients will be divided in two groups. In both groups a verbal and clear detailed information will be given on the intraoperative approach. The first group will receive topical tranexamic acid and the second group topical platelet rich plasma; both in the surgical site. Both groups will be assessed before and after the intervention with laboratory results (hemoglobin, hematocrit levels) and drainage drain.

DETAILED DESCRIPTION:
Total knee replacement (TKR) surgery is one the most common orthopedic procedure in the world. Morbidity in perioperative TKR is associated with: blood loss, pain, infection, wound complications, stiffness, and thrombotic events. Blood loss and transfusion have been associated with an increased hospital stay, costs, morbidity, and mortality. Indications for blood transfusions are now limited and it is well known that is not a free risk procedure. Complications such as; ABO incompatibility, viral transmission, hemolysis, immunosuppression, and wound infection have been reported.

Literature reports have reported blood loss in TKR ranging from 300ml to 1 liter, and transfusion rate varying from 10-38%. In diminishing hospital cost Moskal J. et al. reported 53.90% of savings and a 100% reduction in working hours of the hospital staff using topical tranexamic acid in TKR. Tranexamic acid is an antifibrinolytic agent that acts inhibiting the plasminogen, stabilizing the blood clot; it is used to stop surgical or traumatic bleeding like in the CRASH-2 trial, demonstrating its efficiency in polytraumatized patients. Tranexamic acid has been used in the last years for blood loss with good results. Due to its systemic effects and past medical history of myocardial infarction, stents, and previous thromboembolic events its intravenous use is limited. In this study, the investigators used topical tranexamic acid and its use has been proven in clinical trials as a secure strategy for blood loss reduction in TKR, without excluding patients with previous thromboembolic events.

Platelet-rich plasma (PRP) is an orthobiologic that has played an important role over the past decade in different areas like; spinal fusion, anterior cruciate ligament reconstruction, osteoarthritis, and tendinopathies. The use of PRP in orthopedics is overrated and true indications for its use and cost-benefit are still unclear. Retrospective studies like Pace T et al in 268 patients did not demonstrate differences in-hospital stay, Postoperative hemoglobin levels, and range of motion using PRP in TKR. Morishita M. et al. in a clinical trial of 40 patients, using intralesional PRP didn´t show any benefits for blood loss reduction in TKR, but good clinical results were observed in clinical scores like Knee injury and Osteoarthritis Outcome Score (KOOS) and Visual Analog Scale (VAS) compared to the control group. Other studies have demonstrated the efficacy of topical PRP in blood loss reduction in TKR.

Due to its high platelet concentration and growth factors contained in the alfa granules; it is used as a hemostatic, analgesic, and antiseptic agent in TKR.

There is a variety of blood loss prevention strategies for TKR and these strategies can be divided into preoperative, intraoperative, or postoperative. This study aimed to compare the use of topical tranexamic acid versus topical platelet-rich plasma.

An Insall knee approach, parapatellar medial will be used in all the patients. After the final cuts of the femoral, tibial and patellar and before placing the final cemented components the experimental intervention of the study will begin.

Group 1. A dose of 2 gr of tranexamic acid (1000mg/10 mL X-GEN pharmaceuticals inc.) is diluted in 80 mL of physiologic solution and will be divided into two applications:

First application: 40 mL of the solution previously prepared is applied over the surgical site and it will be left for five minutes then drained out completely by suction.

Second application: The rest of the 40 mL of solution previously prepared is applied after placing the final TKR cemented components (femoral, tibial, and patellar), over the surgical site and leaving it there without draining it by suction.

Group 2. In the preoperative room with previous premedication, a total of 55 mL of total venous blood is obtained from the forearm (cubital o basilic veins). The blood is carried on 12 sterile tubes using sodium citrate at 3.8% (BD, Vacutainer; Becton, Dickinson and Company, NJ). Blood samples are then transported to the Bone and Tissue Bank for centrifugation (1800 rpm for 10 minutes) to separate blood into the 3 layers (White, yellow and red). The superior layer rich in plasma will be collected in 50 microliters polypropylene tubes (Corning, NY). A final volume of 16 ml of platelet-rich plasma is obtained and transferred to airtight tubes (BD Vacutainer; Becton, Dickinson and Company, NJ). The manipulation of the blood samples is made on laminar flow cabin biosecurity class II (Logic 3440801; Labconco, KC). The platelet-rich plasma will be activated with calcium gluconate at 10% (Pisa Farmacéutica, Jalisco, México) before using it is placed in the surgical site topically. The PRP simple will be divided into two applications, initiating the intervention after the final cuts of the TKR components (like the tranexamic acid group).

First application: 8 ml of PRP are applied over the surgical site and are left for five minutes then drained out completely by suction.

Second application: The rest of the 8 ml are applied over the surgical site after placing the final TKR cemented components (femoral, tibial, and patellar), over the surgical site and leaving it without draining.

Then a primary closure of the wound is performed (capsule, fascia, subcutaneous tissue, and skin) in both groups. Close drainage (Drenovac, NEdren S de R.L. de C.V.) is left intraarticular and fixed to the skin. The drainage will be clamped for 2 hours and removed at the 48 hours of the surgery. Thromboprophylaxis (low weight heparin) will be initiated after 6 hours of the end of the surgery. In the postoperative follow-up, any patient with hemoglobin levels less than 9mg/dL with the anemic syndrome will be transfused.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Patient candidates for primary total knee replacement
3. Patients willing to participate in the study and sign de inform consent

Exclusion Criteria:

1. Patients with previous history of thromboembolic event in the last 6 months
2. Patients candidates for revision total knee replacement
3. Patients candidates for tumoral total knee replacement
4. Patients candidates for bilateral total knee replacement
5. Patient with cognitive deficit
6. Previous history of coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09; Primary Completion 2017-03-09 (Actual); Study Completion 2017-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felix Vilchez, MD, PHD, Principal Investigator — Hospital Universitario, Universidad Autonoma de Nuevo Leon
Locations (1):
- Facultad de Medicina UANL, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Levine BR, Haughom B, Strong B, Hellman M, Frank RM. Blood management strategies for total knee arthroplasty. J Am Acad Orthop Surg. 2014 Jun;22(6):361-71. doi: 10.5435/JAAOS-22-06-361. PMID 24860132
- [Background] Wind TC, Barfield WR, Moskal JT. The effect of tranexamic acid on blood loss and transfusion rate in primary total knee arthroplasty. J Arthroplasty. 2013 Aug;28(7):1080-3. doi: 10.1016/j.arth.2012.11.016. Epub 2013 Mar 28. PMID 23541868
- [Background] Frisch NB, Wessell NM, Charters MA, Yu S, Jeffries JJ, Silverton CD. Predictors and complications of blood transfusion in total hip and knee arthroplasty. J Arthroplasty. 2014 Sep;29(9 Suppl):189-92. doi: 10.1016/j.arth.2014.03.048. Epub 2014 May 24. PMID 25007727
- [Background] Moskal JT, Harris RN, Capps SG. Transfusion cost savings with tranexamic acid in primary total knee arthroplasty from 2009 to 2012. J Arthroplasty. 2015 Mar;30(3):365-8. doi: 10.1016/j.arth.2014.10.008. Epub 2014 Oct 12. PMID 25458093
- [Background] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Background] Sheth U, Simunovic N, Klein G, Fu F, Einhorn TA, Schemitsch E, Ayeni OR, Bhandari M. Efficacy of autologous platelet-rich plasma use for orthopaedic indications: a meta-analysis. J Bone Joint Surg Am. 2012 Feb 15;94(4):298-307. doi: 10.2106/JBJS.K.00154. PMID 22241606
- [Background] Patel JN, Spanyer JM, Smith LS, Huang J, Yakkanti MR, Malkani AL. Comparison of intravenous versus topical tranexamic acid in total knee arthroplasty: a prospective randomized study. J Arthroplasty. 2014 Aug;29(8):1528-31. doi: 10.1016/j.arth.2014.03.011. Epub 2014 Mar 21. PMID 24768543
- [Background] Chimento GF, Huff T, Ochsner JL Jr, Meyer M, Brandner L, Babin S. An evaluation of the use of topical tranexamic acid in total knee arthroplasty. J Arthroplasty. 2013 Sep;28(8 Suppl):74-7. doi: 10.1016/j.arth.2013.06.037. PMID 24034510
- [Background] Georgiadis AG, Muh SJ, Silverton CD, Weir RM, Laker MW. A prospective double-blind placebo controlled trial of topical tranexamic acid in total knee arthroplasty. J Arthroplasty. 2013 Sep;28(8 Suppl):78-82. doi: 10.1016/j.arth.2013.03.038. Epub 2013 Jul 29. PMID 23906869
- [Background] Sarzaeem MM, Razi M, Kazemian G, Moghaddam ME, Rasi AM, Karimi M. Comparing efficacy of three methods of tranexamic acid administration in reducing hemoglobin drop following total knee arthroplasty. J Arthroplasty. 2014 Aug;29(8):1521-4. doi: 10.1016/j.arth.2014.02.031. Epub 2014 Mar 6. PMID 24726174
- [Background] Alshryda S, Mason J, Sarda P, Nargol A, Cooke N, Ahmad H, Tang S, Logishetty R, Vaghela M, McPartlin L, Hungin AP. Topical (intra-articular) tranexamic acid reduces blood loss and transfusion rates following total hip replacement: a randomized controlled trial (TRANX-H). J Bone Joint Surg Am. 2013 Nov 6;95(21):1969-74. doi: 10.2106/JBJS.L.00908. PMID 24196467
- [Background] Pace TB, Foret JL, Palmer MJ, Tanner SL, Snider RG. Intraoperative platelet rich plasma usage in total knee arthroplasty: does it help? ISRN Orthop. 2013 Jul 28;2013:740173. doi: 10.1155/2013/740173. eCollection 2013. PMID 24971180
- [Background] Morishita M, Ishida K, Matsumoto T, Kuroda R, Kurosaka M, Tsumura N. Intraoperative platelet-rich plasma does not improve outcomes of total knee arthroplasty. J Arthroplasty. 2014 Dec;29(12):2337-41. doi: 10.1016/j.arth.2014.04.007. Epub 2014 Apr 13. PMID 24851794
- [Background] Aggarwal AK, Shashikanth VS, Marwaha N. Platelet-rich plasma prevents blood loss and pain and enhances early functional outcome after total knee arthroplasty: a prospective randomised controlled study. Int Orthop. 2014 Feb;38(2):387-95. doi: 10.1007/s00264-013-2136-6. Epub 2013 Oct 11. PMID 24114251
- [Background] Bloomfield MR, Klika AK, Molloy RM, Froimson MI, Krebs VE, Barsoum WK. Prospective randomized evaluation of a collagen/thrombin and autologous platelet hemostatic agent during total knee arthroplasty. J Arthroplasty. 2012 May;27(5):695-702. doi: 10.1016/j.arth.2011.09.014. Epub 2011 Oct 27. PMID 22035976
- [Background] Gardner MJ, Demetrakopoulos D, Klepchick PR, Mooar PA. The efficacy of autologous platelet gel in pain control and blood loss in total knee arthroplasty. An analysis of the haemoglobin, narcotic requirement and range of motion. Int Orthop. 2007 Jun;31(3):309-13. doi: 10.1007/s00264-006-0174-z. Epub 2006 Jul 1. PMID 16816947

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 Tranexamic Acid: A dosis of 2 gr of tranexamic acid (1000mg/10ml X-GEN pharmaceuticals inc.) diluted in 80ml of physiologic solution and will be divided in two applications.
  First application: 40ml of the solution previously prepared is applied over the surgical site and it will be left for five minutes then drained out completely by suction.
  Second application: The rest of 40ml of solution previously prepared is applied after placing the final total knee replacement components (femoral, tibial and patellar), over the surgical site and leaving it without draining it by suction.
  Group 1 Tranexamic Acid: 2 gr of tranexamic acid will be applied on the surgical site.
- Group 2 Platelet Rich Plasma: A final volumen of 16 ml of platelet rich plasma is obtained from the forearm vein of the patient and will be divided in two applications.
  First application: 8 mL of Platelet rich plasma are applied over the surgical site and are left for five minutes then drained out completely by suction.
  Second application: The rest of the 8 mL are applied after placing the final TKR cemented components (femoral, tibial and patellar), over the surgical site and leaving it without draining.
  Group 2 Platelet rich plasma: 16ml of platelet rich plasma will be applied of the surgical site
Period: Overall Study
Arm/Group | Group 1 Tranexamic Acid | Group 2 Platelet Rich Plasma
Started | 19 | 21
Baseline | 19 | 21
24 Hours | 19 | 21
48 Hours | 19 | 21
72 Hours | 19 | 21
Completed | 19 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1 Tranexamic Acid: A dosis of 2 gr of tranexamic acid (1000mg/10ml X-GEN pharmaceuticals inc.) diluted in 80ml of physiologic solution and will be divided in two applications.
  First application: 40ml of the solution previously prepared is applied over the surgical site and it will be left for five minutes then drained out completely by suction.
  Second application: The rest of 40ml of solution previously prepared is applied after placing the final TKR components (femoral, tibial and patellar), over the surgical site and leaving it without draining it by suction.
  Group 1 Tranexamic Acid: 2 gr of tranexamic acid will be applied on the surgical site.
- Group 2 Platelet Rich Plasma: A final volumen of 16 ml of platelet rich plasma is obtained from the forearm vein of the patient and will be divided in two applications.
  First application: 8 ml of PRP are applied over the surgical site and are left for five minutes then drained out completely by suction.
  Second application: The rest of the 8 ml are applied after placing the final TKR cemented components (femoral, tibial and patellar), over the surgical site and leaving it without draining.
  Group 2 Platelet rich plasma: 16ml of platelet rich plasma will be applied of the surgical site
- Total: Total of all reporting groups
Arm/Group | Group 1 Tranexamic Acid | Group 2 Platelet Rich Plasma | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (9.3) | 63.8 (6.9) | 66.3175 (8.300478525)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 10 | 9 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Mexico | 19 | 21 | 40
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.9 (3.8) | 31.5 (4.4) | 31.215 (4.033332989)
Overweight [Count of Participants; unit: Participants] | 8 | 8 | 16
Obesity Grade I [Count of Participants; unit: Participants] — Class 1: Body mass index of 30 to < 35
  Participants | 10 | 10 | 20
Obesity Grade II [Count of Participants; unit: Participants] — Class 2: Body mass index of 35 to < 40
  Participants | 0 | 1 | 1
Obesity Grade III [Count of Participants; unit: Participants] — Class 3: Body mass index of 40 or higher. Class 3 obesity is sometimes categorized as "extreme" or "severe" obesity.
  Participants | 1 | 2 | 3
Hemoglobin (g/dL) [Mean (Standard Deviation); unit: g/dL] | 13.6 (1.4) | 13.6 (1.5) | 13.6 (1.416686274)
Hematocrit (% red blood cells) [Mean (Standard Deviation); unit: %] — The proportion of blood that is made up of red blood cells expressed as a percentage or fraction. For example, 40% means 40 milliliters of red blood cells in 100 milliliters of whole blood. The percentage of red blood cells typically represents 37% to 49% of the volume of blood.
  % | 41.6 (4.2) | 41.4 (4.2) | 41.495 (4.094871793)

OUTCOME MEASURES:

1. Primary Outcome: Therapeutic Effect on Hemoglobin Level
Description: The blood test will be taken at 6am every day. Using the same laboratory parameters.
Time Frame: up to 3rd day post operative (Baseline, 24, 48 and 72hrs)
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- Group 2 Platelet Rich Plasma: A final volume of 16 ml of platelet rich plasma is obtained from the forearm vein of the patient and will be divided in two applications.
  First application: 8 ml of PRP are applied over the surgical site and are left for five minutes then drained out completely by suction.
  Second application: The rest of the 8 ml are applied after placing the final TKR cemented components (femoral, tibial and patellar), over the surgical site and leaving it without draining.
  Group 2 Platelet rich plasma: 16ml of platelet rich plasma will be applied of the surgical site
Arm/Group | Group 1 Tranexamic Acid | Group 2 Platelet Rich Plasma
Number analyzed (Participants) | 19 | 21
g/dL
  Baseline | 13.6 (1.4) | 13.6 (1.5)
  24 hours | 10.3 (1.6) | 9.9 (1.1)
  48 hours | 9.5 (1.4) | 9.2 (1.3)
  72 hours | 9.3 (1.5) | 9.1 (1.7)

2. Secondary Outcome: Therapeutic Effect on Hematocrit Level
Description: The blood test will be taken at 6am every day. Using the same laboratory parameters.
Time Frame: up to 3rd day post operative (Baseline, 24, 48 and 72hrs)
Measure: Mean (Standard Deviation); unit: percentage of Hematocrite
Arm/Group | Group 1 Tranexamic Acid | Group 2 Platelet Rich Plasma
Number analyzed (Participants) | 19 | 21
percentage of Hematocrite
  Baseline | 41.7 (4.2) | 41.5 (4.8)
  24 hours | 31.6 (5.0) | 29.8 (3.0)
  48 hours | 29.1 (4.4) | 27.7 (3.3)
  72 hours | 28.6 (4.7) | 27.3 (4.7)

3. Secondary Outcome: Therapeutic Effect on Drainage Quantification
Description: The blood quantification will be taken at 6am every day.
Time Frame: up to 2nd day post operative (24 and 48 hrs)
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Group 1 Tranexamic Acid | Group 2 Platelet Rich Plasma
Number analyzed (Participants) | 19 | 21
mL
  24 hours | 246.4 (152.3) | 263.2 (192.6)
  48 hours | 120.8 (94.6) | 140.2 (127.7)

ADVERSE EVENTS:
Time Frame: up to 3rd day post operative
Arm/Group | Group 1 Tranexamic Acid | Group 2 Platelet Rich Plasma
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 0/19 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/56/NCT02650856/Prot_SAP_000.pdf